CLINICAL TRIAL: NCT01652443
Title: Relationships and Health in the OEF/OIF Veteran Population
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 11-0488
Record Dates: First submitted 2011-12-28; First posted 2012-07-30 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Stress Disorder; Marriage; Suicidal Ideation
Keywords: OEF/OIF Veterans; Relationships
MeSH Terms: conditions — Stress Disorders, Traumatic; Suicidal Ideation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The current study will explore relationships and health in the OEF/OIF Veteran population. Specifically, this study will examine PTSD symptom severity, traumatic brain injury, relationship satisfaction, leisure, general health ratings, feelings of burdensomeness and belongingness, and suicidal ideation.

DETAILED DESCRIPTION:
United States military troops returning home from Operation Enduring Freedom and Operation Iraqi Freedom deployments are presenting with "invisible wounds". These "invisible wounds" include mental health conditions such as posttraumatic stress disorder and traumatic brain injury. Recent literature has begun to explore how PTSD affects the service member, as well as their significant others. Several studies have shown that Veteran endorsement of PTSD symptoms is associated with decreased relationship satisfaction. Prior literature has shown that spending time together and engaging in pleasurable activities as a couple are important strategies for enduring relationship quality and satisfaction. Literature has demonstrated moderate relationships between PTSD and suicidal ideation. A previous study conducted by two of the investigators in this population showed that perceived feelings of burdensomeness and belongingness and identification of suicide as a potential strategy for dealing with these feelings. Joiner has hypothesized that acquired capacity of painful experiences, perceived burdensomeness and thwarted belongingness are the three components of increased suicide risk. Yet few studies exist that examine these constructs in the military population, though research indicates the clinical utility for exploring these constructs and related consequences.

ELIGIBILITY:
Inclusion Criteria:

* OEF/OIF Veteran (at least one OEF/OIF deployment)
* Currently receiving or eligible to receive health care services at DVAMC
* In a current, established relationship for a duration of at least one year
* Age of 18-50

Exclusion Criteria:

* Inability to provide informed consent.
* Inability to adequately respond to questions regarding the informed consent procedure.
* Do not meet the inclusion criteria listed above.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: OEF/OIF Veterans receiving or eligible to receive care at the VA
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Relationship satisfaction | One study visit
  Four item relationship satisfaction survey

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Betthauser, MBA, Principal Investigator — VA VISN 19 MIRECC
Locations (1):
- Eastern Colorado Healthcare System, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: VA VISN 19 MIRECC website — http://www.mirecc.va.gov/visn19/